CLINICAL TRIAL: NCT00107341
Title: A Phase II Trial of PS-341 in Combination With Paclitaxel and Carboplatin for Metastatic Adenocarcinoma of the Lower Esophagus, Gastroesophageal Junction, and Gastric Cardia
Brief Title: Bortezomib, Paclitaxel, and Carboplatin in Treating Patients With Unresectable, Metastatic Cancer of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N044B; NCI-2012-02646 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000413896 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage IV esophageal cancer; recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Bortezomib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bortezomib + paclitaxel + carboplatin (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, and 8 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years.
  Interventions: Drug: bortezomib; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: bortezomib
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with paclitaxel and carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with paclitaxel and carboplatin works in treating patients with unresectable, metastatic cancer of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the confirmed tumor response rate in patients with unresectable, metastatic adenocarcinoma of the esophagus, gastroesophageal junction, or gastric cardia treated with bortezomib, paclitaxel, and carboplatin.

Secondary

* Determine the time to tumor progression, overall survival, and duration of response in patients treated with this regimen.
* Determine the adverse events in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, and 8 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 2. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 25-60 patients will be accrued for this study within 17 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of 1 of the following sites:

  * Esophagus
  * Gastroesophageal junction
  * Gastric cardia

    * No greater than 2 cm from the gastroesophageal junction into the stomach
* Unresectable, metastatic disease
* Not a candidate for potentially curative therapy AND no other more reasonable potentially curative conventional therapy exists
* At least 1 measurable lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 6 months after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No uncontrolled infection
* No chronic debilitating disease
* No prior allergic reaction to carboplatin or paclitaxel
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for recurrent or metastatic disease
* No prior biologic therapy for recurrent or metastatic disease
* No concurrent prophylactic colony-stimulating factors (filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* No prior chemotherapy for recurrent or metastatic disease
* Prior chemotherapy in the neoadjuvant or adjuvant setting (after complete resection of the original tumor) allowed
* Prior combination chemotherapy and radiotherapy allowed provided patient achieved a complete response AND the last dose of combination therapy was administered ≥ 6 months ago

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* No prior radiotherapy for recurrent or metastatic disease
* Prior radiotherapy in the neoadjuvant or adjuvant setting (after complete resection of the original tumor) allowed
* No prior radiotherapy to > 25% of bone marrow for locally advanced disease
* More than 4 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior open abdominal exploration (e.g., laparotomy)
* More than 2 weeks since prior minimally invasive procedures (e.g., laparoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response rate | Up to 3 years

SECONDARY OUTCOMES:
Time to tumor progression | Up to 3 years
Overall survival | Up to 3 years
Duration of response | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Background] Jatoi A, Foster NR, Egner JR, Burch PA, Stella PJ, Rubin J, Dakhil SR, Sargent DJ, Murphy BR, Alberts SR. Older versus younger patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction, and stomach: a pooled analysis of eight consecutive North Central Cancer Treatment Group (NCCTG) trials. Int J Oncol. 2010 Mar;36(3):601-6. doi: 10.3892/ijo_00000535. PMID 20126980
- [Result] Jatoi A, Dakhil SR, Foster NR, Ma C, Rowland KM Jr, Moore DF Jr, Jaslowski AJ, Thomas SP, Hauge MD, Flynn PJ, Stella PJ, Alberts SR. Bortezomib, paclitaxel, and carboplatin as a first-line regimen for patients with metastatic esophageal, gastric, and gastroesophageal cancer: phase II results from the North Central Cancer Treatment Group (N044B). J Thorac Oncol. 2008 May;3(5):516-20. doi: 10.1097/JTO.0b013e31816de276. PMID 18449005